CLINICAL TRIAL: NCT02667236
Title: A Randomized, Double-Blind, Vehicle-Controlled, Parallel Group Study of the Safety and Effectiveness of A-101 Solution 40% in Subjects With Seborrheic Keratosis on the Trunk, Extremities and Face.
Brief Title: A Study of A-101 Solution 40% in Subjects With Seborrheic Keratosis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Aclaris Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A-101-SEBK-301
Record Dates: First submitted 2016-01-26; First posted 2016-01-28 (Estimated); Results first posted 2017-11-13 (Actual); Last update posted 2018-02-06 (Actual); Status verified 2016-12

CONDITIONS: Seborrheic Keratosis
Keywords: seborrheic keratosis
MeSH Terms: conditions — Keratosis, Seborrheic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A-101 Solution (Active Comparator): A-101 Solution 40% administered once
  Interventions: Drug: A-101 Solution
- Vehicle Solution (Placebo Comparator): Vehicle Solution administered once
  Interventions: Other: Vehicle Solution

INTERVENTIONS:
Drug: A-101 Solution — Active Drug
  Arms: A-101 Solution
Other: Vehicle Solution — Placebo
  Arms: Vehicle Solution

SUMMARY:
This is a randomized, double-blind, vehicle-controlled, parallel group study of A-101 Solution 40% compared with Vehicle Solution.

DETAILED DESCRIPTION:
This is a randomized, double-blind, vehicle-controlled, parallel group study. During this study, the investigator will identify 4 eligible SK Target Lesions on each subject on the trunk, extremities and face. The Target Lesions will be treated, by an investigational staff member other than the evaluating investigator, a maximum of two times.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age
2. Clinical diagnosis of stable clinically typical seborrheic keratosis
3. Subject has 4 appropriate seborrheic keratosis Target Lesions on the trunk, extremities and face that each are eligible for treatment as defined below:

   * Have a clinically typical appearance
   * Have a PLA of 2 or greater and be a discrete lesion
   * Not be covered with hair which, in the investigator's opinion, would interfere with the study medication treatment or the study evaluations
   * Not be in an intertriginous fold
   * Not be on the eyelids
   * Not be within 5mm of the orbital rim
   * Not be pedunculated
4. If the subject is a woman of childbearing potential, she has a negative urine pregnancy test and agrees to use an active method of birth control for the duration of the study
5. Subject is non-pregnant and non-lactating
6. Subject is in good general health and free of any known disease state or physical condition which, in the investigator's opinion, might impair evaluation of any Target Lesion or which exposes the subject to an unacceptable risk by study participation
7. Subject is willing and able to follow all study instructions and to attend all study visits
8. Subject is able to comprehend and willing to sign an Informed Consent Form.

Exclusion Criteria:

1. Subject has clinically atypical and - or rapidly growing seborrheic keratosis lesions
2. Subject has presence of multiple eruptive seborrheic keratosis lesions (Sign of Lesser -Trelat)
3. Subject has a current systemic malignancy
4. Subject has used any of the following systemic therapies within the specified period prior to enrollment:

   * Retinoids; 180 days
   * Glucocortico-steroids;
   * Anti-metabolites (e.g., methotrexate);
5. Subject has used any of the following topical therapies within the specified period or in a proximity to any Target Lesion, that in the investigator's opinion interferes with the study medication treatment or the study assessments:

   * LASER, light or other energy based therapy (e.g., intense pulsed light, photo-dynamic therapy;
   * Liquid nitrogen, electrodesiccation, curettage, imiquimod, 5-flurouracil, or ingenol mebutate;
   * Retinoids;
   * Microdermabrasion or superficial chemical peels;
   * Glucocortico-steroids or antibiotics
6. Subject currently has or has had any of the following within the specified period or in a proximity to any Target Lesion that, in the investigator's opinion, interferes with the study medication treatment or the study assessments:

   * A cutaneous malignancy;
   * A sunburn; currently
   * A pre-malignancy (e.g., actinic keratosis); currently
   * Body art (e.g., tattoos, piercing, etc.); currently
   * Excessive tan; currently
7. Subject has a history of sensitivity to any of the ingredients in the study medications
8. Subject has any current skin disease (e.g., psoriasis, atopic dermatitis, eczema, sun damage, etc.), or condition (e.g., sunburn, excessive hair, open wounds) that, in the opinion of the investigator, might put the subject at undue risk by study participation or interfere with the study conduct or evaluations
9. Subject has participated in an investigational drug trial in which administration of an investigational study medication occurred within 30 days prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Actual)
Dates: Start 2016-01; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stuart D Shanler, MD, Study Director — Chief SCience Officer
Locations (1):
- Aclaris Therapeutics, Inc., Malvern, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Smith SR, Xu S, Estes E, Shanler SD. Anatomic Site-Specific Treatment Response With 40% Hydrogen Peroxide (w/w) Topical Formulation for Raised Seborrheic Keratoses: Pooled Analysis of Data from Two Phase 3 Studies. J Drugs Dermatol. 2018 Oct 1;17(10):1092-1098. PMID 30365590

RESULTS

PARTICIPANT FLOW:
Groups:
- A-101 Solution: A-101 Solution 40% applied topically
  A-101 Solution: Active Drug
- Vehicle Solution: Vehicle Solution applied topically
  Vehicle Solution: Placebo
Period: Overall Study
Arm/Group | A-101 Solution | Vehicle Solution
Started | 223 | 227
Completed | 220 | 226
Not Completed | 3 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | A-101 Solution | Vehicle Solution | Total
Number analyzed (Participants) | 223 | 227 | 450
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 72 | 55 | 127
  >=65 years | 151 | 172 | 323
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (8.42) | 69.1 (8.71) | 68.7 (8.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 126 | 264
  Male | 85 | 101 | 186
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 214 | 216 | 430
  Unknown or Not Reported | 4 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 4 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 219 | 221 | 440
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 223 | 227 | 450

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects With Target Lesion Clearance as Assessed by the Physician Lesion Assessment
Description: Proportion of subjects for whom all target lesions were judged to be clear on the Physician Lesion Assessment Scale (PLA=0) at Visit 8. The PLA Scale is a 4 point scale used by the investigator to assess each subject's target SK Lesion.
Time Frame: Day 106 of the study
Population: ITT Population; all randomized subjects
Measure: Count of Participants; unit: Participants
Arm/Group | A-101 Solution | Vehicle Solution
Number analyzed (Participants) | 223 | 227
Participants | 9 | 0

2. Secondary Outcome: Proportion of Subjects With 3 of 4 Target Lesion Clearance
Description: Proportion of Subjects for whom at least 3 of 4 target lesions were judged to be clear on the Physician Lesion Assessment (PLA=0) at Visit 8
Time Frame: Day 106 of the study
Population: ITT population; all randomized subjects
Measure: Count of Participants; unit: Participants
Arm/Group | A-101 Solution | Vehicle Solution
Number analyzed (Participants) | 223 | 227
Participants | 30 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected from V2 (Day 1) through V8 (Day 106)
Arm/Group | A-101 Solution | Vehicle Solution
All-Cause Mortality (participants affected / at risk) | 0/223 | 0/227
Serious Adverse Events (participants affected / at risk) | 4/223 | 6/227
Other Adverse Events (participants affected / at risk) | 10/223 | 14/227
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A-101 Solution (N=223) | Vehicle Solution (N=227)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Gastric Ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Central nervous system lesion (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 1 (1)
Mental Status Changes (Psychiatric disorders) | 0 (0) | 1 (1)
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A-101 Solution (N=223) | Vehicle Solution (N=227)
Nasopharyngitis (Infections and infestations) | 3 (3) | 7 (7)
Bronchitis (Infections and infestations) | 3 (3) | 1 (1)
Upper Respiratory Infection (Infections and infestations) | 1 (1) | 3 (3)
Actinic Keratosis (Skin and subcutaneous tissue disorders) | 3 (3) | 0 (0)
Seasonal Allergy (Immune system disorders) | 0 (0) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Institution and Investigator agree not to publish the results of this study without the prior written consent of Sponsor.